CLINICAL TRIAL: NCT03913949
Title: A Phase I Study of the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics Properties of Orally Administered APG-2575 in Patients With Hematologic Malignancies
Brief Title: A Study to Evaluate the Safety,PK and PD of APG-2575 in Patients With Hematologic Malignancies
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Ascentage Pharma Group Inc. (Industry)
Collaborators: Suzhou Yasheng Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: APG-2575-CN-001
Record Dates: First submitted 2019-04-10; First posted 2019-04-12 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Chronic Lymphocytic Leukemia; Non Hodgkin Lymphoma
Keywords: APG-2575; B-cell lymphoma 2 (BCL-2); Chronic lymphocytic leukemia; non-hodgkin's lymphoma
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, Non-Hodgkin | interventions — Lisaftoclax

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- single-agent, open-label, Phase I study of APG-2575 (Experimental): The study consists of the dose escalation stage and the dose expansion stage
  Interventions: Drug: APG-2575

INTERVENTIONS:
Drug: APG-2575 — Multiple dose cohorts, PO, every day (QD) of a 28-day cycle

SUMMARY:
The purpose of this study is to assess the safety, tolerability, pharmacokinetic and pharmacodynamic properties of APG-2575 in patients with relapse or refractory chronic lymphocytic leukemia and non-hodgkin's lymphoma.

DETAILED DESCRIPTION:
This is a multi-center, single-agent, open-label, Phase I study of APG-2575. The study consists of the dose escalation stage and the dose expansion stage. APG-2575 will be administered orally, once daily for consecutive 4 weeks as one cycle. Initially, the start dose is 20mg. Single patient cohorts will be evaluated, the dose of APG-2575 will be increased in subsequent cohorts, to 50 mg, 100 mg, 200 mg, 400 mg, 600mg and 800mg accordingly. If there is any one of the following event is observed, a dose-limiting toxicity (DLT), two drug related Grade 2 toxicities or one drug related ≥ Grade 3 toxicity, or laboratory or clinical tumor lysis syndrome (TLS), or suspected hypersensitivity reaction occur in Cycle 1, the dose escalation will convert to the standard 3+3 design, If ≥ 2/6 patients develop DLT at any dose level dose escalation will cease and the dose level immediately below will be expanded to 6 patients. If ≤ 1/6 patients develop a DLT at the highest dose reached this will be declared the MTD. After the MTD/Recommended Phase II Dose (RP2D) is defined, a maximum of 40 patients will be treated at that dose level.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years old.
2. Histologically confirmed diagnosis of chronic lymphocytic leukemia, or non-Hodgkin's lymphoma such as mantle cell lymphoma, diffuse large B cell lymphoma, Waldenstrom macroglobulinemia (WM).
3. Patient must have relapsed or refractory to, intolerant to, or are considered ineligible for therapies known to provide clinical benefit.
4. Life expectancy ≥ 3 months.
5. Eastern Cooperative Oncology Group (ECOG) Performance Status (PS): 0 -1 in dose escalation; 0-2 in dose expansion.
6. Corrected QT interval ≤450ms in males, and ≤470ms in females.
7. Adequate bone marrow function independent of growth factor:

   1. Absolute neutrophil count (ANC) ≥1.0 X 10E9/L.
   2. Hemoglobin ≥ 8.0 g/dL.
   3. Platelets count ≥ 30 X 10E9/L (entry platelet count must be independent of transfusion within 7 days of first dose).
8. Adequate renal and liver function as indicated by:

   1. Serum creatinine ≤ 1.5 x upper limit of normal (ULN); if serum creatinine is >1.5 X ULN, creatinine clearance must be ≥60 mL/min.
   2. Total bilirubin ≤1.5 x ULN, except subject with known Gilbert's syndrome.
   3. Aspartate aminotransferase (AST) and Alanine aminotransferase (ALT) <2.5 x ULN.
   4. Alkaline phosphatase < 2.5 x ULN and < 5 x for bone metastases &/or no hepatic parenchymal metastases on screening radiographic examination.
   5. Thromboplastin time (aPTT)≤1.5 X ULN unless the subject is receiving anticoagulant therapy as long as prothrombin time (PT) or aPTT is within therapeutic range of intended use of anticoagulants.
9. Willingness by both males, and female patients of child bearing potential, to use contraception by a method that is deemed effective by the investigator, throughout the treatment period and for at least three months following the last dose of study drug Postmenopausal women must be amenorrheal for at least 12 months to be considered of non-childbearing potential. All partners must have the same willingness for contraception methods throughout the treatment period and for at least three months following the last dose of study drug as well.
10. Ability to understand and willingness to sign a written informed consent form (the consent form must be signed by the patient prior to any study-specific procedures).
11. Willingness and ability to comply with study procedures and follow-up examination.

Exclusion Criteria:

Patients who meet any of the following exclusion criteria are not to be enrolled in this study:

1. Prior history of allogeneic cell transplant.
2. Subjects have been diagnosed with Burkitt's lymphoma, Burkitt-like lymphoma, or lymphoblastic lymphoma/leukemia.
3. Received chemotherapy within 14 days prior to entering the study.
4. Received biologic (< 28 days), small molecule targeted therapies (< 5 half-life) or other anti-cancer therapy within 21 days of study entry.
5. Concurrent treatment with an investigational agent, 14 days for small molecular agents and/or 28 days for biologics treatment prior to the first dose of therapy.
6. Radiation within 14 days of study entry, thoracic radiation within 28 days of study entry.
7. Has gastrointestinal conditions that could affect the absorption of APG-2575 in the opinion of the Investigator.
8. Has known active central nervous system (CNS) involvement.
9. Continuance of toxicities due to prior radiotherapy or chemotherapy agents that do not recover to ≤ Grade 1 except alopecia or neuropathy.
10. Failure to recover adequately, as judged by the investigator, from prior surgical procedures. Patients with active wound healing, patients who have had major surgery within 28 days from study entry, and patients who have had minor surgery within 14 days of study entry.
11. Unstable angina, myocardial infarction, or a coronary revascularization procedure within 180 days of study entry.
12. Active rheumatoid arthritis (RA), active inflammatory bowel disease, or any other disease or condition associated with chronic inflammation.
13. Active infection requiring systemic antibiotic/ antifungal medication, known clinically active hepatitis B or C infection, or known HIV disease.
14. Known or suspected Wilson's Disease, or other conditions that affect copper accumulation or regulation.
15. Uncontrolled concurrent illness including, but not limited to: symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with the study requirements.
16. The last treatment for the subject before signing the informed consent was bcl-2 targeted drug treatment (if the subject had received bcl-2 inhibitor treatment but did not develop drug resistance, it could be included in this study).
17. History of secondary active malignancies within the past 2 years. However, adequately treated superficial skin cancer other than melanoma, in-situ cervix cancer more than 4 weeks, or prostate cancer not requiring any treatment and under surveillance prior to enrollment will not be considered exclusionary.
18. Known to be allergic to study drug ingredients or their analogues.
19. Pregnancy or lactation, or pregnancy is expected during the study period or within 3 months after the last administration of APG-2575.
20. Any other condition or circumstance that would, in the opinion of the investigator, make the patient unsuitable for participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Estimated)
Dates: Start 2019-06-03 (Actual); Primary Completion 2024-10-20 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) | 28 days
  Patients with APG-2575 treatment related adverse events (AE), serious adverse events (SAE) will be assessed according NCI CTCAE Version 5.0

SECONDARY OUTCOMES:
Maximum plasma concentration (Cmax) | 28 days
  Maximum plasma concentration (Cmax) will be assessed in the patients treated with APG-2575
Area under the plasma concentration versus time curve (AUC) | 28 days
  Area under the plasma concentration versus time curve (AUC) of APG-2575 will be assessed in the patients treated with APG-2575
Anti-tumor effects of APG-2575 | up to 3 years
  Response will be evaluated every 2 cycles (8 weeks), by the investigator based on disease specific criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Jianxiang Wang, MD, Principal Investigator — Blood Diseases Hospital Chinese Academy of Medical Sciences
Locations (5):
- China (5):
  - Anhui Procincial hospital, Hefei, Anhui
  - Henan Provincial Oncology Hospital, Zhengzhou, Henan
  - Zhongnan Hospital of Wuhan University, Wuhan, Hubei
  - Blood Diseases Hospital Chinese Academy of Medical Sciences, Tianjin, Tianjin Municipality
  - The First Affiliated Hospital, Zhejiang University School of Medicin, Hangzhou, Zhejiang